CLINICAL TRIAL: NCT05194696
Title: The Impact of Caffeine Consumption on Preventing Cataract
Brief Title: Caffeine Consumption and Cataract Prevention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: CaffQuest
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: Cataract; Caffeine
MeSH Terms: conditions — Cataract | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caffeine questionnaire: A questionnaire concerning caffeine habits will be handed out to the patients
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Patients have to answer a questionnaire about their caffeine consumption habits during lifetime

SUMMARY:
Effect of peroral caffeine consumption on the delay of cataract onset.

DETAILED DESCRIPTION:
Several experimental studies have shown that caffeine inhibits cataract development by scavenging reactive oxygen species. Evidence from epidemiological studies, however, is controversial. Varma et al., found that the incidence of cataract blindness in humans was significantly lower in groups consuming higher amounts of coffee in comparison to the groups with lower coffee intake. Moreover, Rautiainen et al. showed that the dietary total antioxidant capacity including coffee of middle-aged and elderly women was inversely associated with the risk of age-dependent cataract. Another population-based study involving the population residing in Beaver Dam, Wisconsin, did not find a meaningful association between 10-year cumulative incidence of cataract and the amount of caffeine intake.

Although cataracts can be surgically removed, barriers that prevent access to surgery are a problem in many countries. Moreover, no prophylactic treatments are currently available to prevent the onset of cataract. Yet estimates indicate that a delay of only 10 years in the onset of cataract could reduce the need for cataract surgery by as much as 50%.

The present study aims to investigate whether peroral caffeine consumption on a regular daily basis for a significant period of time and sufficient dose delays cataract development.

12000 eyes of 6000 patients will be included into this study. Patient will have to fill out a questionnaire for caffeine consumption habits during lifetime and risk factors for cataract development. Further, a complete ophthalmic examination, cataract grading, refraction, visual testing, and biometry will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age older than 21 years
* cataract

Exclusion Criteria:

- age younger than 21 years

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cataracts awaiting cataract surgery
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Caffeine consumption | 48 months
  Caffeine consumption will be assessed using a questionnaire concerning the caffeine drinking habits

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No